CLINICAL TRIAL: NCT05619796
Title: Assessment of Clinical and Radiographic Efficiency of Manual and Pediatric Rotary File Systems in Primary Root Canal Preparation
Brief Title: Assessment of Clinical & Radiographic Efficiency of Manual & Pediatric Rotary Systems in Primary Root Canal Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shaimaa Shaban Mohamed El-desouky, Lecturer of Pediatric dentistry, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #R-PED-9-22-2
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Manual; Rotation; Obturation; Post Operative Pain
Keywords: Cone-beam computed tomography; kedo-S square; Fanta AF™ Baby
MeSH Terms: conditions — Bites and Stings; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A randomized, controlled prospective clinical study
Who Masked: Participant, Outcomes Assessor
Masking Description: the quality of root canal filling by two trained pediatric dentists, blinded to instrumentation technique.
  A nursing officer who was blind to the study groups, had trained all parents on how to record the postoperative pain.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1: Kedo-S Square rotary files (Experimental): Primary root canals(n=20) were instrumented using rotary P1 Kedo-S Square files (Reeganz Dental Care Pvt. Ltd. India) at 300 rpm and 2.2N cm torque. The rotary files were used with an Endo-Mate DT endodontic motor (NSK, Tokyo, Japan) and EDTA gel 17% (Meta Biomed Co. Ltd, Chungbuk, Korea) was used before instrumentation.
  Interventions: Procedure: pulpectomy procedure; Radiation: Post-operative Cone Beam Computed Tomography; Other: Post-operative pain assessment
- group II: Fanta AFTM-Baby rotary system (Experimental): Primary root canals(n=20) were instrumented using Fanta AFTM-Baby rotary system (Shanghai Fanta Dental Materials, SUNGO Certification Company Limited, London, England) at 350 rpm and 2 N cm torque. Four files were used sequentially in the following order; open file #17/0.08, #20/0.04 yellow, #25/0.04 red and #30/0.04 blue. The rotary files were used with an Endo-Mate DT endodontic motor (NSK, Tokyo, Japan) and EDTA gel 17% (Meta Biomed Co. Ltd, Chungbuk, Korea) was used before instrumentation.
  Interventions: Procedure: pulpectomy procedure; Radiation: Post-operative Cone Beam Computed Tomography; Other: Post-operative pain assessment
- group III: manual K-files (Active Comparator): Primary root canals(n=20) were instrumented using No.15 till 35 size manual K-files (Mani, Inc, Japan) using the quarter-turn-pull technique.
  Interventions: Procedure: pulpectomy procedure; Radiation: Post-operative Cone Beam Computed Tomography; Other: Post-operative pain assessment

INTERVENTIONS:
Procedure: pulpectomy procedure — single visit pulpectomy was performed under strict aseptic conditions by a single operator. Peri-operative evaluation was done using intraoral digital senso. The teeth were anesthetized with 2% mepivacaine with 1:20,000 levonordefrin & isolated using rubber dam. caries was removed using no. 330 round carbide burs in high-speed contra angle headpiece. Access opening was gained & the roof of the pulp chamber was removed. Working length was determined by apex locator, then confirmed by periapical radiograph. Working length will be determined 1 mm shorter than apex. mechanical preparation was done using the tested files according to each group. Then, canals were irrigated with 1% sodium hypochlorite between each file followed by irrigation with normal saline. The root canals were dried using paper points & root canals were filled with Metapex. Intermediate restorative material was placed, and the tooth was restored with a preformed stainless-steel crown in the same appointment.
Radiation: Post-operative Cone Beam Computed Tomography — post-operative CBCT image was taken after completing the procedure with fixed exposure parameters (120 Kv, 5mA and 0.125mm voxel size) using smallest field of view (8D, 8Hcm) to improve spatial resolution. The CBCT images were obtained by using 3D module of On Demand Dental software (version 1.0 (build 1.0.10.7462),× 64 Edition, copyright 2004-2017 Cybermed, Korea and license key 670094709).
  The Immediate post-operative CBCT was taken to evaluate the quality of root canal filling by two trained pediatric dentists, blinded to instrumentation technique .
  Other Names: Obturation Quality Assessment
Other: Post-operative pain assessment — The parents of the children were given a questionnaire to record the intensity of postoperative pain at six, twelve, twenty-four and forty-eight hours after the pulpectomy procedure. A nursing officer who was blind to the study groups, had trained all parents on how to record the postoperative pain. The four-point pain intensity scale was used to record postoperative pain (figure 5). This scale categorizes pain as follows: (1) no pain; (2) slight pain; (3) moderate pain; and (4) severe pain. To ensure standardization, the same parent was asked to record the child's pain intensity at all time intervals. To reduce the possibility of the parents failing to record the pain at a given time, the investigator also recorded findings via telephonic conversation with the parents. The children returned to the department two days after the pulpectomy procedure with their completed questionnaire form.

SUMMARY:
Manual files used for the pulpectomy of primary teeth have some disadvantages such as time wastage and the occurrence of iatrogenic errors compared to rotary systems.

Little studies have been done to clinically evaluate the Kedo-S Square & Fanta AF™ Baby rotary systems in relation to the quality of obturation, instrumentation time and postoperative pain in root canal preparation of primary molars using CBCT.

DETAILED DESCRIPTION:
Biomechanical preparation is one of the most important steps of primary teeth pulpectomy, which are primarily targeted during canal debridement . Conventionally, hand files were used for cleaning and shaping in primary teeth with some disadvantages such as time wastage and the occurrence of iatrogenic errors such as zipping, lateral perforations, apical obstruction, and canal transportation.

The use of rotary instruments for primary tooth instrumentation is faster, affordable, and yields consistent, reliable results. Numerous rotary endodontic systems designed primarily for application in permanent teeth, have been suggested for primary teeth root canal preparation. Since the primary teeth have a ribbon-shaped anatomy and shorter, thinner curved roots than permanent teeth, the use of these files in pulpectomy of primary teeth could produce lateral perforations. As a result, there was a great need for the development of a unique pediatric rotary file system.

The Kedo-S Square rotary system is a single file system specifically designed for paediatric use. It consists of two files, one for anterior primary teeth (A1) and one for posterior primary teeth (P1) also, Fanta AF™-Baby rotary system, another specifically generated paediatric rotary file, was produced using Ni-Ti controlled memory (CM)-Wire technology.

A good root canal treatment in primary teeth is dependent on the quality of biomechanical preparation, the type of obturating material used with as few voids as possible, and the achievement of a good hermetic seal. Also, treatment time is an important aspect as reduced chairside time increases children's cooperation for dental treatment, reduces anxiety, and making the treatment protocol optimal. Another factor affecting the success of primary teeth pulpectomy is the postoperative pain which may be due to extrusion of foreign particles into peri-radicular tissues accordingly, causing inflammation and releasing inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* healthy cooperative children
* non-vital posterior teeth with sufficient coronal structure
* intact 2/3rd root structure
* no mobility or external pathological root resorption

Exclusion Criteria:

* Uncooperative children
* children with systemic illness
* non-restorable primary molars
* primary molars with sever mobility, or pathological root resorption

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-09-04 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Root canal preparation using Manual and Pediatric Rotary File Systems during pulpectomy of primary teeth | 2 days
  by evaluation of the obturation quality using immediate post-operative CBCT which is assessed by two trained pediatric dentists, blinded to instrumentation technique .
  The quality of obturation was assessed by evaluating the length of the Metapex filling according to Coll and Sadrian criteria :
  * Under filling (Score 1): Canal filled with metapex more than 2 mm short of the apex.
  * Optimal filling (Score 2): Canal filling ending at the radiographic apex or up to 2 mm short of apex.
  * Overfilling (Score 3): Any canal showing filling outside the root apex.

SECONDARY OUTCOMES:
postoperative pain after primary teeth pulpectomy using Manual and Pediatric Rotary File Systems | 2 days
  using four-point pain intensity scale. This scale categorizes pain as follows: (1) no pain; (2) slight pain; (3) moderate pain; and (4) severe pain.
  The parents of the children were given a questionnaire to record the intensity of postoperative pain at six, twelve, twenty-four and forty-eight hours after the pulpectomy procedure.
  A nursing officer who was blind to the study groups, had trained all parents on how to record the postoperative pain.
  To ensure standardization, the same parent was asked to record the child's pain intensity at all time intervals.
  To reduce the possibility of the parents failing to record the pain at a given time, the investigator also recorded findings via telephonic conversation with the parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Barr ES, Kleier DJ, Barr NV. Use of nickel-titanium rotary files for root canal preparation in primary teeth. Pediatr Dent. 2000 Jan-Feb;22(1):77-8. PMID 10730297
- [Background] Jeevanandan G, Govindaraju L. Clinical comparison of Kedo-S paediatric rotary files vs manual instrumentation for root canal preparation in primary molars: a double blinded randomised clinical trial. Eur Arch Paediatr Dent. 2018 Aug;19(4):273-278. doi: 10.1007/s40368-018-0356-6. Epub 2018 Jul 12. PMID 30003514
- [Background] Mohamed RH, Abdelrahman AM, Sharaf AA. Evaluation of rotary file system (Kedo-S-Square) in root canal preparation of primary anterior teeth using cone beam computed tomography (CBCT)-in vitro study. BMC Oral Health. 2022 Jan 18;22(1):13. doi: 10.1186/s12903-021-02021-0. PMID 35042489
- [Background] Abd El Fatah YAM, Khattab NMA, Gomaa YF, Elheeny AAH. Cone-beam computed tomography analysis of primary root canals transportation and dentin loss after instrumentation with two-pediatric rotary files. BMC Oral Health. 2022 May 31;22(1):214. doi: 10.1186/s12903-022-02245-8. PMID 35641977
- [Background] Elheeny AAH, Abdelmotelb MA. Postoperative pain after primary molar pulpectomy using rotary or reciprocating single files: A superior, parallel, randomized clinical trial. Int J Paediatr Dent. 2022 Nov;32(6):819-827. doi: 10.1111/ipd.12959. Epub 2022 May 5. PMID 35152509